CLINICAL TRIAL: NCT03635437
Title: A Phase I/II, 3-Arm, Open Label, Single Centre Study to Investigate the Safety and Effect of Oral GABA Therapy on Beta-Cell Regeneration in Type 1-diabetes Patients
Brief Title: Evaluation of Safety and Diabetes Status Upon Oral Treatment With GABA in Patients With Longstanding Type-1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Per-Ola Carlsson (Other)
Collaborators: Diamyd Medical AB (Industry)
Responsible Party: Sponsor-Investigator, Per-Ola Carlsson, Professor, Senior consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Regenerate-1 (G/P2/18/1)
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Remygen; GABA
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gamma-Aminobutyric Acid; Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose gamma-aminobutyric acid (GABA) (Experimental): Oral GABA treatment 200 mg daily for 6 months
  Interventions: Drug: Gamma-Aminobutyric Acid (GABA)
- High dose gamma-aminobutyric acid (GABA) (Experimental): Oral GABA treatment 600 mg daily for 6 months
  Interventions: Drug: Gamma-Aminobutyric Acid (GABA)
- High dose gamma-aminobutyric acid (GABA) + Alprazolam (Experimental): Oral Alprazolam treatment 0.5 mg daily combined with oral GABA treatment 600 mg daily for 3 months. Alprazolam treatment thereafter ended, and study subjects will continue with oral GABA treatment 600 mg daily only for another 3 months.
  Interventions: Drug: Gamma-Aminobutyric Acid (GABA); Drug: Alprazolam

INTERVENTIONS:
Drug: Gamma-Aminobutyric Acid (GABA) — Patients eligible for the main study will be randomized in a 1:1:1 ratio stratified by the C-peptide level to receive 200 mg of GABA (Remygen) for 6 months, 600 mg of GABA (Remygen) for 6 months, or Alprazolam 0.5 mg combined with GABA 600 mg (Remygen) for 3 months followed by treatment with GABA 600 mg (Remygen) only for another 3 months. The start of the arms with high dose GABA will be delayed and started first after that a data safety monitoring board has evaluated and approved the safety data of the first 4 patients included in the arm with low dose GABA. All patients will continue to receive intensive insulin treatment from their personal physicians during the whole study period.
  Other Names: GABA (Remygen)
Drug: Alprazolam — Patients eligible for the main study will be randomized in a 1:1:1 ratio stratified by the C-peptide level to receive 200 mg of GABA (Remygen) for 6 months, 600 mg of GABA (Remygen) for 6 months, or Alprazolam 0.5 mg combined with GABA 600 mg (Remygen) for 3 months followed by treatment with GABA 600 mg (Remygen) only for another 3 months. The start of the arms with high dose GABA will be delayed and started first after that a data safety monitoring board has evaluated and approved the safety data of the first 4 patients included in the arm with low dose GABA. All patients will continue to receive intensive insulin treatment from their personal physicians during the whole study period.
  Arms: High dose gamma-aminobutyric acid (GABA) + Alprazolam

SUMMARY:
The main goal of this study is to find a reasonably safe and tolerable treatment for adult patients with type 1-diabetes and that regain some of the endogenous insulin secretion, improve the patients' quality of life (QoL) and reduce the risk of both short- and long-term complications. The hypothesis tested is that oral GABA treatment with the newly developed compound Remygen will be safe and induce regain of some endogenous insulin secretion in adult patients with type 1-diabetes diagnosis for more than five years. The first part of the study will include 6 patients and be performed as a Safety and Dose Escalation study in three steps. The main study is a three-arm, open label, single center, clinical trial. Eligible patients will be randomized into one of three active treatment arms to receive oral GABA treatment for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given by patients according to national regulations
2. Type 1 diabetes diagnosed ≥ 5 years at the time of screening
3. Must have been diagnosed with Type 1-diabetes before the age of 25
4. Age ≥18 and ≤50
5. Fasting c-peptide levels should be in the range from not detectable levels up to <0.12 nmol/L
6. For males of childbearing potential adequate contraception is as follows:

   1. condom (male)
   2. abstinence from heterosexual intercourse
   3. female partner using contraception as below listed:

      * oral (except low-dose gestagen (lynestrenol and norethisterone)), injectable, or implanted hormonal contraceptives
      * combined (estrogen and progestogen containing)
      * oral, intravaginal or transdermal progesterone hormonal contraception associated with inhibition of ovulation
      * intrauterine device
      * intrauterine hormone-releasing system (for example, progestin-releasing coil)
      * bilateral tubal occlusion

Exclusion Criteria:

1. Females of child-bearing potential
2. Previous or current treatment with immunosuppressant therapy (although topical and inhalation steroids are accepted)
3. Treatment with any oral or injected anti-diabetic medications other than insulin
4. Patients on medications which may disturb GABA action, such as Baclofen, Valium, Acamprosate, Neurontin, or Lyrica
5. HbA1c > 90 mmol/mol
6. eGFR <60 ml/min
7. Increased plasma concentrations of alanine aminotransferase (>0.75 μkatl/l for females or >1.1 μkat/l for males) and/or aspartate aminotransferase (>0.60 μkat/l for females or >0.75μkat/l for males).
8. Known cancer disease
9. Known sleeping apnea or pulmonary disorder with carbon dioxide rentention in blood
10. Previous history of pancreatitis or other exocrine pancreatic disorder
11. A history of epilepsy, myasthenia gravis, head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles
12. A history of alcohol or drug abuse
13. A significant illness other than diabetes within 2 weeks prior to first dosing
14. Known human immunodeficiency virus (HIV) or hepatitis
15. Females who are breastfeeding
16. Males not willing to use adequate contraception during the study period.
17. Known hypersensitivity agains benzodiazepins or any excipients of study drugs
18. Participation in other clinical trials with a new chemical entity within 3 months or 5 half-lives of the new chemical entity, whatever longest.
19. Inability or unwillingness to comply with the provisions of this protocol
20. Deemed by the investigator not being able to follow instructions and/or follow the study protocol or other reasons that, at the investigator's discretion, could affect the subject's current clinical condition during study procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Adverse events possibly or probably related to GABA treatment | 6 months
  To evaluate the acute and long-term safety of oral GABA treatment. The endpoint will investigate number of adverse events possibly or probably related to GABA treatment.

SECONDARY OUTCOMES:
Difference in C-peptide response to mixed meal tolerance test before and directly after treatment | 6 months
  Difference in C-peptide (Area under the curve 0-120 min) during a mixed meal tolerance test between baseline and after 6 months of oral GABA treatment
Difference in C-peptide response to mixed meal tolerance test during and after treatment | 7 months
  Difference in C-peptide (Area under the curve 0-120 min) during a mixed meal tolerance test between baseline and after 3 and and 6 months of treatment and between baseline and the follow-up visit
Difference in maximum stimulated C-peptide to mixed meal tolerance test during and after treatment | 7 months
  Difference in maximum stimulated C-peptide during a mixed meal tolerance test between baseline and after 3 and 6 months of treatment and between baseline and the follow-up visit.
Difference in C-peptide response to mixed meal tolerance test during and after treatment between treatment groups | 7 months
  Difference in C-peptide (Area under the curve 0-120 min) during a mixed meal tolerance test between treatment group 1 and 2 and after 3 and 6 months of treatment and between baseline and the follow-up visit
Difference in glucagon response during a hypoglycemic clamp before and after treatment | 7 months
  Difference in glucagon (area under the curve) during a hypoglycemic clamp between baseline and 6 months of treatment
Difference in glucagon response during a hypoglycemic clamp between treatment groups before and after treatment | 7 months
  Difference in glucagon (area under the curve) during a hypoglycemic clamp between treatment group 1 and 2 between baseline and 6 months of treatment
Change in HbA1c by treatment | 7 months
  Change in HbA1c between 0,3 and 6 months of treatment and at the follow-up one month later.
Change in exogenous insulin consumption by treatment | 7 months
  Change in exogenous insulin consumption between 0,3 and 6 months of treatment and at the follow-up one month later.
Change in fasting C-peptide by treatment | 7 months
  Change in fasting C-peptide levels between 0,3 and 6 months of treatment and at the follow-up one month later.
Change in variables that indicate effects on immune system | 7 months
  Change by treatment in variables that indicate effects on the immune system such as serum autoantibodies to GAD65 and islet antigen-2, and immune cells
Change in GABA plasma levels | 7 months
  Analysis of GABA plasma levels after 0, 3 and 6 months of treatment and at the follow-up visit one month later.
Change in diabetes treatment satisfaction questionnaire | 7 months
  Measurements of patient diabetes treatment satisfaction by questionnaire during study. Each of eight questions have a 7-graded scale from 0-6. 48 points are therefore maximal treatment satisfaction and comparisons will be made to score before treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Espes D, Liljeback H, Hill H, Elksnis A, Caballero-Corbalan J, Carlsson PO. GABA induces a hormonal counter-regulatory response in subjects with long-standing type 1 diabetes. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002442. doi: 10.1136/bmjdrc-2021-002442. PMID 34635547